CLINICAL TRIAL: NCT04496817
Title: Effects of DHA and Lutein Enriched Eggs on Retina Health and Metabolic and Physical Parameters in Type 2 Diabetes: a Strategy for Diabetic Retinopathy
Brief Title: Enriched Eggs for Retina Health in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Egg Farmers of Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B2020:007
Record Dates: First submitted 2020-07-24; First posted 2020-08-03 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Retinopathy; Type 2 Diabetes
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 2 | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled, parallel trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enriched Egg Group (Experimental): Participants will consume 2 medium sized docosahexaenoic acid and lutein enriched eggs daily (at least 5 days per week) for 6 weeks.
  Interventions: Other: Docosahexaenoic Acid and Lutein Enriched Eggs
- Regular Egg Group (Placebo Comparator): Participants will consume 2 medium sized non-enriched eggs daily (at least 5 days per week) for 6 weeks.
  Interventions: Other: Regular Eggs

INTERVENTIONS:
Other: Docosahexaenoic Acid and Lutein Enriched Eggs — Consumption of 2 docosahexaenoic acid and lutein enriched eggs daily (at least 5 days our week) for 6 weeks
  Arms: Enriched Egg Group
Other: Regular Eggs — Consumption of 2 non enriched eggs daily (at least 5 days our week) for 6 weeks
  Arms: Regular Egg Group

SUMMARY:
Diabetes mellitus has been declared a major public health issue. Among the complications of the disease, retinopathy can have a significant impact on mobility and quality of life for individuals living with diabetes. As the leading cause of new blindness in adults, diabetic retinopathy has been shown to affect 23% of all Type 1 and 14% of Type 2 diabetic individuals. Various studies have reported that a number of components in the egg may contribute to visual function and eye health. Specifically, i) egg yolk naturally contains, and can be further enriched with the carotenoids lutein and zeaxanthin. Lutein and zeaxanthin protect the retina against light induced retinal damage by acting as potent antioxidants that shield the retina from harmful short-wave radiation. ii) eggs can also be enriched to provide a vehicle for specific nutrients to promote eye health including omega-3 fatty acid, docosahexaenoic acid (DHA). A substantial amount of DHA is uniquely found within the retina. A DHA deficiency has shown to induce abnormal retina function indicating a constant supply of this nutrient is necessary for retina health. Currently, the American Diabetes Association declares that eggs are an excellent choice for people with diabetes, but information lacks on the status of whole egg consumption in diabetic individuals in relation to their retinal health. Therefore, the current study aims to determine if the consumption of two lutein and DHA enriched eggs per day can safely improve the retina function of individuals with type 2 diabetes.

A total of 60 adult diabetic male and female participants will be recruited to take part in this double-blinded, randomized, placebo-controlled, parallel trial. Participants will be randomly assigned to include two DHA and lutein enriched eggs or regular eggs into their usual diet for 6 weeks. At the beginning and end of the trial, a variety of measures will be analyzed including blood lipid parameters, carotenoid status, anthropometrics, arterial stiffness, advanced glycated end products, macular pigment optical density and electroretinography. These measures will aid in determining whether enriched egg consumption can safely improve retina function, while not adversely effecting body composition and cardiovascular risk factors in individuals with diabetes. The results of this study will contribute to the development of valuable prevention strategies for eye health in individuals with diabetes, thereby improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>19 years of age)
* Individuals diagnosed with Type 2 diabetes
* Individuals taking oral hypoglycemic medications (sulfonylureas, meglitinides, biguanides, thiazolidinediones etc.)
* Individuals with a fasting plasma glucose of ≥7.0 mmol/L or glycated hemoglobin (A1C) of ≥6.5%. (these values are based on the Canadian Diabetes Association and are predictors of the development of diabetic retinopathy)

Exclusion Criteria:

* Individuals previously diagnosed with moderate to severe diabetic retinopathy (to assess egg consumption as a preventative strategy for diabetic retinopathy).
* Individuals with eye disease (cataracts, glaucoma, age-related macular degeneration, retinitis pigmentosa, optic atrophy, and eye malformation etc.)
* Individuals with Alzheimer's, dementia or other mental cognitive diseases
* Individuals with Type 1 diabetes
* Individuals taking insulin
* Individuals diagnosed with cancer or anemia
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Retina Function | 6 weeks
  Measured by Full Field Electroretinography

CONTACTS AND LOCATIONS:
Overall Officials: Miyoung Suh, RD, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Asper Clinical Research Institute, Winnipeg, Manitoba, Canada